CLINICAL TRIAL: NCT03155477
Title: Effect Of Curcuma Xanthorrhiza Supplementation In Systemic Lupus Erythematosus Patients (SLE) With Hypovitamin D Which Were Given Vitamin D3 Towards Disease Activity (SLEDAI), Interleukin-6 (IL-6) And Tumor Growth Factor-β1 (TGF-β1) Serum
Brief Title: Effect Of Curcuma Xanthorrhiza and Vitamin D3 Supplementation in SLE Patients With Hypovitamin D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saiful Anwar Hospital (Other)
Responsible Party: Principal Investigator, Cameleia Diah Setyorini, Medical Doctor, Saiful Anwar Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01/2016/SLE/CurcuminvitaminD
Record Dates: First submitted 2017-05-13; First posted 2017-05-16 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: SLE
Keywords: SLE, vitamin D, SLEDAI, IL-6, TGF- β1
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Cholecalciferol" and "C. Xanthorrhiza" (Experimental): Subjects received Cholecalciferol 400 IU 3 times daily and C. Xanthorrhiza 20 mg 3 times daily per oral for 3 months (group II, n=19)
  Interventions: Dietary Supplement: "Cholecalciferol" and "C. Xanthorrhiza"
- "Cholecalciferol" and "placebo" (Placebo Comparator): Subjects received cholecalciferol 3×400 IU and placebo 3×1 tablet for 3 months (group I, n=20).
  Interventions: Dietary Supplement: "Cholecalciferol" and "placebo"

INTERVENTIONS:
Dietary Supplement: "Cholecalciferol" and "C. Xanthorrhiza" — Cholecalciferol are given 400 IU 3 times daily for 3 months C. Xanthorrhiza are given 200 mg 3 times daily for 3 months
  Other Names: Teorol 400 IU Novell Pharmaceutical Laboratories; Curcuma Soho Industries Pharmacy
  Arms: "Cholecalciferol" and "C. Xanthorrhiza"
Dietary Supplement: "Cholecalciferol" and "placebo" — Cholecalciferol are given 400 IU 3 times daily for 3 months Placebo are given 3 times daily for 3 months
  Other Names: Teorol 400 IU Novell Pharmaceutical Laboratories
  Arms: "Cholecalciferol" and "placebo"

SUMMARY:
This a double blind randomised controlled trial (RCT) to determine the effect of Curcuma Xanthorrhiza supplementation on vitamin D3 administration to disease activity (SLEDAI), IL-6 and TGF-β1 serum in SLE patients with hypovitamin D. SLE patients with hypovitamin D had milder disease activity, lower IL-6 and higher TGF-β1 serum level when supplemented with Curcuma Xanthorrhiza and vitamin D3 compared with vitamin D3 and placebo.

DETAILED DESCRIPTION:
Cholecalciferol 1200 IU supplementation for 3 months in hypovitamin D SLE patients, decrease SLEDAI, however, it has not reached the mild activity and remission yet. Curcumin contained in Curcuma Xanthorrhiza; is an immunomodulator that has similar biological effect with vitamin D. Combination of curcumin and vitamin D are expected to work synergistically.

The subjects who fulfilled inclusion criteria, willing to participate in the research and signed the informed consent were 40 patients. Research subjects were randomized using simple randomization. The subjects were divided into 2 groups: the group receiving 3×400 IU cholecalciferol and 3×1 tablet placebo (group I, n=20), and the group receiving 3×400 IU and curcumin (Curcuma Xanthorrhiza) 3x20 mg for 3 months (group II, n=20).

Fifteen cc of venous blood samples were taken for complete blood tests, liver function (SGOT/SGPT), renal function (ureum/creatinine), vitamin D (25(OH)D), calcium, anti-dsDNA, C3, C4, IL-6 and serum TGF-β1. Examination of vitamin D levels using Enzyme Immuno Assay method (Diasorin Inc, Stillwater, MN USA), anti-dsDNA levels using ELISA (Bioluminescenassay), C3, C4, IL-6 and serum TGF-β1 using ELISA (Biolegend). Proteinuria was examined using a urine spot sample while with enzymatic-turbidimetric methods. SLE disease activity was assessed using SLEDAI score. Laboratory and SLEDAI examination were performed at the beginning of the study and the end of the study; except for the serum calcium levels examined each month to determine the side effects of the drug.

Patients continue to receive the usual immunosuppressive drugs (corticosteroids, chloroquine, cyclophosphamide, mycophenolate mofetil, azathioprine, and cyclosporine), as well as calcium, antihypertensive drugs and other routine medications. Regular drugs, cholecalciferol, Curcuma Xanthorrhiza and placebo, are administered by a physician in the Rheumatology Outpatient Clinic who is not a member of the research team in different examination rooms.

The results are presented in mean ± standard deviation, median (IQR 25-75%) and n (%). The homogeneity test of variance using Levene. The Saphiro-Wilk test is used to determine the normality of the data, assuming the normality of the data is fulfilled if p> 0.05. Different tests after treatment in both study groups used a non-paired/Mann-Whitney test. The influence between variables was tested using Spearman/Pearson correlation test. Data analysis uses Statistical Package for the Social Sciences Software version 22 (SPSS Inc, Chicago IL). Differences and correlations are said to be significant when the value of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* SLE based on the criteria of American Collage of Rheumatology (ACR) 1997
* Active SLE (SLEDAI> 3)
* 25(OH)D level <30 ng/ml.

Exclusion Criteria:

* Pregnant
* Taking supplements containing vitamin D and cur cumin
* Had liver function disorders (SGOT/SGPT levels> 2.5 times the upper normal limit)
* Had impaired renal function (GFR <25 ml/min)
* Severe infections such as tuberculosis, pneumonia or HIV

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
SLE disease activity | 3 months
  SLE disease activity was assessed using SLEDAI in the last 10 days

SECONDARY OUTCOMES:
IL-6 | 3 months
  IL-6 serum level (pg/ml)
TGF-β1 | 3 months
  TGF-β1 serum level (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Handono Kalim, Prof., Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Handono K, Pratama MZ, Endharti AT, Kalim H. Treatment of low doses curcumin could modulate Th17/Treg balance specifically on CD4+ T cell cultures of systemic lupus erythematosus patients. Cent Eur J Immunol. 2015;40(4):461-9. doi: 10.5114/ceji.2015.56970. Epub 2016 Jan 15. PMID 26862311
- [Derived] Singgih Wahono C, Diah Setyorini C, Kalim H, Nurdiana N, Handono K. Effect of Curcuma xanthorrhiza Supplementation on Systemic Lupus Erythematosus Patients with Hypovitamin D Which Were Given Vitamin D3 towards Disease Activity (SLEDAI), IL-6, and TGF-beta1 Serum. Int J Rheumatol. 2017;2017:7687053. doi: 10.1155/2017/7687053. Epub 2017 Dec 28. PMID 29445400